CLINICAL TRIAL: NCT00003139
Title: A Phase III Study to Test the Efficacy of the Prophylactic Use of Oral Pilocarpine to Reduce Hyposalivation and Mucositis Associated With Curative Radiation Therapy in Head and Neck Cancer Patients
Brief Title: Pilocarpine in Preventing Mucositis and Dry Mouth in Patients Receiving Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: RTOG-9709; CDR0000065912; NCI-P97-0121
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Head and Neck Cancer; Oral Complications
Keywords: oral complications; lip and oral cavity squamous cell carcinoma; oropharyngeal squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphoid Interstitial Pneumonia; Squamous Cell Carcinoma of Head and Neck | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pilocarpine hydrocloride (Experimental): 5mg pilocarpine hydrochloride tablets commencing 3 days prior to irradiation
  Interventions: Drug: pilocarpine hydrochloride
- Placebo (Placebo Comparator): Placebo tablets commencing 3 days prior to irradiation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: pilocarpine hydrochloride — 5mg pilocarpine hydrochloride tablets
  Arms: Pilocarpine hydrocloride
Other: Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as pilocarpine may protect normal cells from the side effects of radiation therapy. It is not yet known if pilocarpine may be effective in preventing mucositis and dry mouth in patients receiving radiation therapy for head and neck cancer.

PURPOSE: Randomized, double-blinded, phase III trial to study the effectiveness of pilocarpine in preventing mucositis and dry mouth in patients receiving radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether prophylactic use of pilocarpine can shelter unstimulated and stimulated whole salivary flow in patients with head and neck cancer. II. Determine whether prophylactic use of pilocarpine can moderate xerostomia in these patients. III. Determine whether prophylactic use of pilocarpine can reduce the grade and duration of radiation induced mucositis in these patients. IV. Evaluate quality of life outcomes between patients receiving pilocarpine versus placebo. V. Evaluate the impact of xerostomia on patients receiving irradiation to the head and neck.

OUTLINE: This is a randomized, double blind study. Patients receive a central axis midplane dose of radiotherapy five days per week over 6 to 7 weeks. Oral pilocarpine or placebo is administered beginning 3 days prior to radiotherapy, one tablet four times per day for three months. A tablet will be taken 45-60 minutes before radiotherapy. After three months, and after a 3-4 day rest period, all patients receive non blinded pilocarpine for an additional three month period. Patients are followed at weeks 4, 13, and 26 after the start of radiotherapy.

PROJECTED ACCRUAL: A total of 244 patients will be accrued (122 per treatment arm).

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven oral cavity and/or oropharyngeal squamous cell carcinoma Radiation volume to encompass at least 50% of parotid glands and have at least 50 Gy delivered to that volume via external beam No salivary gland malignancies or diseases

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: Karnofsky 60-100% Life Expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Effective contraceptive method must be used during study No pilocarpine allergy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to head or neck Surgery: Not specified Other: No concurrent adrenergic antagonists, cholinergic drugs, anti-cholinergics, or tricyclics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 1998-03; Primary Completion 2001-01 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Acute salivary gland toxicity | From the start of treatment to 13 weeks

SECONDARY OUTCOMES:
Acute mucositis in the pharynx, palate, tongue, or buccal | From the start of treatment to 13 weeks
Quality of life as measured by the University of Washington Head and Neck Symptom questionnaire | Pretreatment to 26 weeks from the start of treatment
Effects of continuing pilocarpine out to 6 months from the start of treatment | From the start of treatment to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francis G. LeVeque, DDS, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (232):
- United States (216):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Urology Associates - Mobile AL, Mobile, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscallosa, Alabama
  - Providence Cancer Therapy Center, Anchorage, Alaska
  - Arizona Cancer Center, Tucson, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Medical Center, Concord, California
  - Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Cancer Care Center, Pomona, California
  - Mercy Medical Center - Redding, Redding, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Santa Cruz Radiation Oncology Medical Group, Inc., Santa Cruz, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University, Stanford, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Radiation Oncology Center - Walnut Creek, Walnut Creek, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Whittingham Cancer Center, Norwalk, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - West Florida Cancer Institute - Pensacola, Pensacola, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - InterCommunity Cancer Center at Rome, Rome, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - St. Joseph's Radiation Oncology Center, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Medical Center at Bowling Green, Bowling Green, Kentucky
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Western Baptist Hospital, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Joint Center for Radiation Therapy, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Ozarks Regional, Springfield, Missouri
  - Veterans Affairs Medical Center - Saint Louis, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Elizabeth General Medical Center - West, Elizabeth, New Jersey
  - South Jersey Hospital - Millville, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - Genesee Hospital - Rochester, Rochester, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - UNI-MED Medical Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - Samaritan Regional Cancer Center, Corvallis, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Penn State Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Catholic Medical Center, Mercy Fitzgerald Divison, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Virginia Baptist Hospital, Lynchburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Swedish Hospital Tumor Institute, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Oncology Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
- Canada (16):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Scarantino C, LeVeque F, Swann RS, White R, Schulsinger A, Hodson DI, Meredith R, Foote R, Brachman D, Lee N. Effect of pilocarpine during radiation therapy: results of RTOG 97-09, a phase III randomized study in head and neck cancer patients. J Support Oncol. 2006 May;4(5):252-8. PMID 16724649
- [Result] Fisher J, Scott C, Scarantino CW, Leveque FG, White RL, Rotman M, Hodson DI, Meredith RF, Foote R, Bachman DG, Lee N. Phase III quality-of-life study results: impact on patients' quality of life to reducing xerostomia after radiotherapy for head-and-neck cancer--RTOG 97-09. Int J Radiat Oncol Biol Phys. 2003 Jul 1;56(3):832-6. doi: 10.1016/s0360-3016(03)00121-4. PMID 12788192
- [Result] Fisher JJ, Scott CB, Scarantino CW, et al.: Phase III quality of life (Qol) study: reduction in hyposalivation does not improve Qol for head and neck (H&N) cancer patients post radiation therapy (P-RT). RTOG 9709. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1423, 2002.
- [Result] Scarantino CW, Leveque FG, Scott CB, et al.: A phase III study of concomitant oral pilocarpine to reduce hypo-salivation and mucositis associated with curative radiation therapy (RT) in the head and neck (H&N) cancer patients. RTOG 9709. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-897, 225a, 2001.
- [Result] Scarantino CW, Leveque F, Scott C, et al.: A phase III study on the concurrent use of oral pilocarpine to reduce hyposalivation and mucositis associated with radiation therapy in head and neck cancer patients: final results of RTOG 97-09. [Abstract] Int J Radiat Oncol Biol Phys 51(3 suppl 1): A-157, 85-86, 2001.